CLINICAL TRIAL: NCT01317251
Title: Effect of Milk and Cheese on Fecal Fat Excretion and Blood Lipid
Acronym: MOFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Mette Kristensen, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: B281
Record Dates: First submitted 2011-03-11; First posted 2011-03-17 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2011-03

CONDITIONS: Obesity
Keywords: Obesity prevention; appetite regulation; hyperlipidemia
MeSH Terms: conditions — Obesity; Hyperlipidemias | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control diet (Experimental): Diet without dairy products
  Interventions: Other: Dietary intervention (without dairy products)
- Milk diet (Experimental): Diet with a high content of milk
  Interventions: Other: Dietary intervention (high milk content)
- Cheese diet (Experimental): Diet with a high content of cheese
  Interventions: Other: Dietary intervention (high cheese content)

INTERVENTIONS:
Other: Dietary intervention (without dairy products) — Control diet without dairy products
  Arms: Control diet
Other: Dietary intervention (high milk content) — Diet with a high content of milk (~1200 mg Ca/d from milk)
  Arms: Milk diet
Other: Dietary intervention (high cheese content) — Diet with a high content of cheese (~1200 mg Ca/d from cheese)
  Arms: Cheese diet

SUMMARY:
The aim is to study the effect of milk versus cheese on fecal fat excretion and blood lipids. To do this, a randomized crossover intervention study with 3 14-day periods (control diet, milk diet, cheese diet) will be conducted in 16 young males. Fasting blood samples will be collected before and after each period, and fecal samples will be collected for the last 5 days in each period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* BMI 20-28 mg/m2

Exclusion Criteria:

* Smoking
* Medicine use
* Dietary supplements
* Lactose intolerance, milk allergy
* Dislike of dairy products
* Excessive physical activity (> 10h/wk)
* Known chronic illnesses

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Fecal fat excretion | During day 10-14 in each period
  Total excretion of fecal fat (grams/day)avaraged over five days

SECONDARY OUTCOMES:
Total, HDL and LDL cholesterol | Day 1 and 14 in each period
Triglycerides | Day 1 and 14 in each period
Appetite sensation | Assessed on day 1, 8 and 14 in each period

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Dr med, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Human Nutrition, University of Copenhagen, Frederiksberg C, Denmark

REFERENCES:
- [Derived] Soerensen KV, Thorning TK, Astrup A, Kristensen M, Lorenzen JK. Effect of dairy calcium from cheese and milk on fecal fat excretion, blood lipids, and appetite in young men. Am J Clin Nutr. 2014 May;99(5):984-91. doi: 10.3945/ajcn.113.077735. Epub 2014 Mar 12. PMID 24622806